CLINICAL TRIAL: NCT00268970
Title: Phase 2 Trial of First-Line Therapy With Satraplatin and Paclitaxel in Patients With Unresectable Stage III or IV Non-small Cell Lung Cancer (NSCLC)
Brief Title: Satraplatin and Paclitaxel in Patients With Advanced Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Agennix (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAT2-05-05
Record Dates: First submitted 2005-12-22; First posted 2005-12-23 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Advanced non-small cell lung cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — satraplatin; Paclitaxel

INTERVENTIONS:
Drug: Satraplatin in combination with Paclitaxel — Paclitaxel 200 mg/m2 IV over 3 hours on day 1. Satraplatin 60 mg/m2 administered by mouth once daily for 5 consecutive days (days 1-5). Satraplatin will be administered within 2 hours following paclitaxel infusion on day 1. Subsequent doses on days 2-5 will be taken at approximately 24 hour intervals.

SUMMARY:
The purpose of this trial is to study the combination regimen of satraplatin and paclitaxel in the first-line treatment of patients with advanced non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
This trial is designed to study the efficacy and safety of a novel oral platinum analog, satraplatin, in combination with another chemotherapy drug, paclitaxel, for the first line of treatment (patients who have not received chemotherapy for disease that has metastasized) of patients with advanced NSCLC.

WHAT IS SATRAPLATIN:

Satraplatin is a member of the platinum-based class of chemotherapy drugs. Platinum-based drugs have been clinically proven to be one of the most effective classes of anticancer therapies. Unlike the currently marketed platinum-based drugs, satraplatin can be given orally.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced NSCLC
* Patients must not have received any prior antineoplastic chemotherapy or investigational product for lung cancer prior to study entry.
* Patients must have at least one unidimensionally measurable lesion definable by magnetic resonance imaging (MRI) or computed tomography (CT) scan.
* ECOG performance status of ≤ 2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-12; Primary Completion 2007-04 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
To examine overall response rates in patients with advanced NSCLC treated with a first-line regimen of satraplatin and paclitaxel | 3 months

SECONDARY OUTCOMES:
To examine time to tumor progression, overall survival, and safety in patients with advanced NSCLC treated with a first-line regimen of satraplatin and paclitaxel | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sarah Cannon Research Institute, Nashville, Tennessee, United States